CLINICAL TRIAL: NCT04249219
Title: Young Adults Responses to E-Cigarette Advertisement Features and the Effect of Restricting Features on Tobacco Use
Brief Title: Responses to E-Cigarette Advertising
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elise Stevens, Assistant Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H00022646; K99DA046563 (NIH)
Record Dates: First submitted 2020-01-24; First posted 2020-01-30 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: E-Cig Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-Cigarette Ads (Experimental): All individuals in the study will see the same e-cigarette advertisements presented in a random order.
  Interventions: Other: Viewing e-cigarette ads

INTERVENTIONS:
Other: Viewing e-cigarette ads — All participants will see the same e-cigarette ads presented in a random order.

SUMMARY:
While conventional cigarette use continues to decline among youth and young adults, e-cigarette (EC) use is on the rise. The use of ECs during young adulthood, particularly 18 years of age, is especially alarming because it is not only a critical period in development but also a time when tobacco use is established. Additionally, the tobacco industry targets individuals of this age with the hope that they will one day progress to using combustible cigarettes. Advertising may be one of the reasons leading young people to use ECs, and the Food and Drug Administration (FDA) now has the authority to regulate EC advertisement features. The goal of the study is to determine which EC ad features most strongly influence young adults' attitudes, susceptibility, and intentions to use ECs. Fifteen ads from the most popular EC brands that employ a brand, product descriptions, and modeling features were selected. Young adults who are susceptible to EC use will come into the lab and view these ads. During exposure, they will be assessed for real-time visual attention using eye-tracking, orienting responses using heart rate, and arousal using skin conductance as well as pre- and post-ad self-report measures of attitudes, susceptibility, and behavioral intentions. These factors will help determine the most high impact features, which will be associated with the greatest visual attention, orienting responses, and arousal levels and changes in attitudes. Findings from this study will provide public health officials important and urgently needed information as to what advertising features are contributing to the sharp rise in the use of ECs among young adults.

ELIGIBILITY:
Inclusion Criteria:

* 18-26 years old,
* Fluent in English,
* Biochemically confirmed abstinence combusted tobacco or marijuana (eCO: exhaled carbon monoxide <6 parts per million) at time of visit
* Reporting never trying an e-cigarette, not even a puff OR reporting having used an e-cigarette in the past but has not used in the past 30 days
* Susceptibility to EC use, will be determined using the Susceptibility to Use Tobacco Products questionnaire

Exclusion Criteria:

* Younger than 18 years or older than 26 years
* Not fluent in English
* Not confirmed abstinent of combusted tobacco or marijuana
* Use of an e-cigarette
* Not susceptible to e-cigarette use

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise M Stevens, PhD, Principal Investigator — UMass Medical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were assigned to the one arm of the study.
Period: Overall Study
Arm/Group | E-Cigarette Ads
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | E-Cigarette Ads
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 62
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (2.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 38
  More than one race | 5
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Attention to Specific ad Feature
Description: Heart rate was measured to assess the cognitive resources allocated to the message. Using three sensors applied to participants' fingers, electrocardiogram (ECG) signals were recorded with a Shimmer 3 EXG module, while viewing the advertisements and were sampled at 512 Hz. Heart change scores were computed using beats per minute (BPM) and subtracting the first second of the stimuli (participant had seen a black screen just prior) from scores for each second of message exposure for each participant. Then, scores were averaged across each advertisement. Lesser values indicated greater deceleration in heart rate, signaling more cognitive resources allocated to the message.
Time Frame: Change from the first second of viewing to each subsequent second of the intervention (10 seconds per ad), averaged for each participant.
Population: All individuals in the study saw the same advertisements.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | E-Cigarette Ads
Number analyzed (Participants) | 62
Beats per minute
  Blu ads | -1.7062 (1.318833535)
  Juul ads | -0.9676 (0.918885902)
  MarkTen ads | -1.8238 (1.209606837)

2. Primary Outcome: Arousal
Description: Skin conductance or galvanic skin response was measured using three sensors applied to participants' fingers. Skin conductance measured if there was an emotional response and the intensity of the emotional response. A "peak" is a biological indicator that something happened, and the participant had an emotional response to it. The amplitude of each peak for each participant was measured and averaged per ad.
Time Frame: The average amplitude of skin conductance peaks over the 10 second viewing window for each ad brand.
Population: All individuals in the study saw the same e-cigarette advertisements.
Measure: Mean (Standard Deviation); unit: microSiemens
Arm/Group | E-Cigarette Ads
Number analyzed (Participants) | 62
microSiemens
  Blu ads | 0.094441599 (0.039786446)
  Juul ads | 0.080156704 (0.014821968)
  MarkTen ads | 0.107337121 (0.047972698)

3. Primary Outcome: Attention to Specific ad Feature
Description: Visual attention was assessed using an eye-tracker connected to the base of the computer screen. For each message, four areas of interest (AOI) were identified: 1) brand, 2) descriptor, 3) modeling, and 4) warning. All four AOIs were summed for a total number of milliseconds that a participant viewed the AOIs.
Time Frame: Duration of seconds spent on all areas of interest during 10 second viewing window for each ad brand
Population: All individuals in the study saw the same e-cigarette advertisements.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | E-Cigarette Ads
Number analyzed (Participants) | 62
milliseconds
  Blu ads | 5464.656 (557.5287713)
  Juul ads | 5963.704 (676.8965371)
  MarkTen ads | 5107.014 (394.2662056)

4. Secondary Outcome: Motivations to Avoid E-cigarettes
Description: Self-report Please rate on a scale from 0 (not at all) to 10 (very much). "How important is it to avoid e-cigarettes in the future?" "How confident are in avoiding e-cigarettes in the future?" "How ready are you to avoid e-cigarettes in the future?" "How committed are you to avoid e-cigarettes in the future?"
  Scores were averaged for each ad for each participant. Then, an overall average was taken among all participants for each ad. Higher values indicate greater motivation to avoid e-cigarettes.
Time Frame: Immediately after viewing each ad
Population: All individuals in the study saw the same e-cigarette advertisements.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-Cigarette Ads
Number analyzed (Participants) | 62
score on a scale
  Blu ads | 8.618 (0.027748874)
  Juul ads | 8.62 (0.051961524)
  MarkTen ads | 8.61 (0)

ADVERSE EVENTS:
Time Frame: The specific period of time over which adverse event data were collected was between the beginning of the participant's visit and the end. The time frame for each participant was one hour and 30 minutes.
Arm/Group | E-Cigarette Ads
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT04249219/Prot_SAP_000.pdf